CLINICAL TRIAL: NCT02599610
Title: Effects of Digital Vaginal Examination During Labor on Pain and Anxiety : a Randomised Controlled Trial
Brief Title: Effects of Digital Vaginal Examination During Labor on Pain and Anxiety Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Erkan Kalafat, Research Assistant, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 006
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Pregnancy; Obstetric Labor
Keywords: labor, vaginal examination, transperineal ultrasound, pain, anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digital vaginal examination (Active Comparator): Patients assigned to this group will be followed-up with digital vaginal examinations as described in intervention protocol.
  Interventions: Other: Digital vaginal examination
- Transperineal ultrasound examination (Experimental): Patients assigned to this group will be followed-up with transperineal ultrasound examinations as described in intervention protocol.
  Interventions: Device: Transperineal ultrasound examination

INTERVENTIONS:
Other: Digital vaginal examination — Patients will be subject to digital vaginal examinations every four hours during latent phase of first stage, hourly during active phase of first stage and as needed during second stage.
  Arms: Digital vaginal examination
Device: Transperineal ultrasound examination — Patients will be subject to transperineal ultrasound examinations every four hours during latent phase of first stage, hourly during active phase of first stage and as needed during second stage.
  Arms: Transperineal ultrasound examination

SUMMARY:
Digital vaginal examination is the most common method for assessing progress of labor and delivery. Considering it is the most common intervention women receive during course of labor, evidence for psychological effects of digital vaginal examination on women is surprisingly sparse. Reducing the number of vaginal examination during labor has been proposed by many authors as benefit of more vaginal examination is unclear. However this is unlikely to happen until more research on the topic demonstrates clear detrimental effects of vaginal examination.

Our study is aimed at investigating association of vaginal examination with psychological distress of women during labor. Anxiety during labor is associated with longer labor duration, increased perception of pain, problems with newborn attachment, and increased rates of postpartum depression and post-traumatic stress disorder. In this study, women were assigned to either digital vaginal examination or transperineal ultrasound assessment groups were compared to each other in a randomised controlled setting.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous women
* Spontaneous active labor
* Cephalic presentation

Exclusion Criteria:

* Women with known psychiatric disorders
* Labor induction
* Advanced labor during admission (Dilatation greater than 7cm)
* Presence of a prenatally diagnosed anomaly in fetus
* Admission to neonatal intensive care unit after delivery
* Delayed hospital discharge due to excessive weight loss of neonate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Anxiety levels | Between 12 to 48 hours
  Anxiety levels of the patients will be assessed with the State-Trait Anxiety Inventory (STAI) questionnaire during admission, at the beginning of active phase of stage one and four hours after delivery.
Labor pain | Between 12 to 48 hours
  Perceived pain level of the patients will be assessed with Visual Analog Scale (VAS) questionnaire during admission, at the beginning of active phase of stage one and four hours after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Erkan Kalafat, MD, Principal Investigator — Ankara University
Locations (1):
- Ankara University Faculty of Medicine, Department of Obstetrics and Gynecology, Ankara, Turkey (Türkiye)